CLINICAL TRIAL: NCT04189718
Title: A Clinical and Radiological Comparison of Osseodensification Versus Conventional Implant Site Preparation Protocol During Dental Implant Placement. A Randomised Controlled Clinical Trial
Brief Title: Comparative Evaluation of Osseodensification Versus Conventional Implant Site
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Principal Investigator, Dr Prabhuji MLV, Professor, Krishnadevaraya College of Dental Sciences & Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_80824
Record Dates: First submitted 2019-12-02; First posted 2019-12-06 (Actual); Last update posted 2019-12-06 (Actual); Status verified 2019-12

CONDITIONS: Bone Density; Implant Stability
Keywords: hounsfield

STUDY DESIGN:
Intervention Model Description: wo groups were made one test and control. The control group were treated with conventional implant site preparation technique and the test group were treated with osseodensification technique.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osseodensification protocol (Experimental): Experimental: In the test group, osteotomy site preparation was performed using Osseodensification technique at 1100 rpm and implant was placed
  Interventions: Procedure: osseodensification protocol; Procedure: conventional implant site preparation protocol
- conventional implant site preparation protocol (Active Comparator): Control: in the control group, osteotomy site was prepared using conventional drilling protocol at 1100 rpm and implant was placed.
  Interventions: Procedure: osseodensification protocol; Procedure: conventional implant site preparation protocol

INTERVENTIONS:
Procedure: osseodensification protocol — Local anaesthesia was administered and mucoperiosteal flap was reflected. Implant osteotomies was performed with sequential drilling with osseodensification protocol at 1100 rpm. The pilot drill was used in clockwise direction and the other sequential drills were used in counter clockwise direction under copious irrigation. Flap closure was achieved using 3-0 silk sutures to protect the implant site.
  Other Names: Densah bur protocol; Osseodensification technique
Procedure: conventional implant site preparation protocol — Local anaesthesia was administered and mucoperiosteal flap was reflected. Implant osteotomies was performed with sequential drilling with conventional implant site preparation protocol at 1100 rpm. The pilot drill was used in clockwise direction and the other sequential drills were used in clockwise direction under copious irrigation. Flap closure was achieved using 3-0 silk sutures to protect the implant site.
  Other Names: standard drilling technique, regular drilling technique

SUMMARY:
The present study is a human, prospective, randomised controlled clinical trial conducted to explore and compare the clinical and radiological outcome of Osseodensification protocol with conventional implant site preparation protocol. The trial is in accordance with the Consolidated Standards of Reporting Trials (CONSORT) criteria, 2010.

DETAILED DESCRIPTION:
Twenty two dental implants were placed in twelve healthy individuals satisfying the inclusion and exclusion criteria were recruited for the study. A detailed, thorough medical and dental history was obtained and each patient was subjected to comprehensive clinical and radiological examination. All patients were informed about the nature of the study, the surgical procedure involved, potential benefits and risks associated with the surgical procedure and written informed consent were obtained from all patients.

All the patients received Norris implant. the implant site preparation technique being Osseodensification protocol for the test group and conventional implant site preparation protocol for the control group, eleven in each group. The clinical and radiographic parameters were recorded at baseline, immediate post implant placement, six months and twelve months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Single/multiple missing teeth in the maxillary anterior/posterior region.
2. Bone density of D2 or D3 (Carl E.Misch).
3. Patients between 18-75 years.
4. Patients who demonstrate good plaque control (PI<10%) and showing good compliance.
5. Patients willing to participate in the study.

Exclusion Criteria:-

1. Insufficient density or height of residual ridge.
2. Patients with bleeding disorder or on anticoagulant therapy.
3. Pregnant and lactating females.
4. Patients with history of smoking.
5. Use of systemic antibiotics in the past 3 months.
6. Patients treated with any medication known to cause periodontal changes.
7. Drug and alcohol abuse.
8. Occlusal interferences.
9. Patients with history of titanium allergy.
10. Immunocompromised state and debilitating disease.
11. Malignancy or radiotherapy/chemotherapy for malignancy.
12. Systemic diseases that would negatively influence wound healing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
primary implant stability | immediate post implant placement
  the primary implant stability was measured during implant placement using Insertion Torque Value(ITV).
change from baseline in bone density | 1 year
  A Multislice CT was used for scanning the implant site pre operatively, just after implant placement and 1 year post implant placement to measure the change in bone density. It was performed using a tube voltage of 120 kV(kilovolt) and a tube current of 40 mA(milliampere). The occlusal plane of the patient was set perpendicular to the floor base using ear rods. The axial images was reconstructed with 0.625 mm thick slices at 0.625 mm interval and a 1.75 mm field of view(FOV) image analysis software
change from baseline in crestal bone level | 1 year
  Digital radiographs (radiovisiograph-RVG) were standardised using radiographic paralleling technique and positioning device and custom fabricated bite-block at baseline and follow up.Mesial and distal peri-implant radiographic bone level were recorded in millimetres on the digital radiographs using Digimiser image

SECONDARY OUTCOMES:
change from baseline in keratinized mucosa width | 1 year
  The width of keratinized mucosa was measured from the mucosal margin to the mucogingival junction at the facial surface. The mucogingival junction location was determined using a visual method (Schiller's potassium iodide solution).
change from baseline in ridge width | 1 year
  Soft tissue and hard tissue labio-lingual ridge width was measured at baseline, immediate post implant placement, 6 months and 1 year after implant placement using ridge mapping calipers/Multislice CT.
Patient reported pain evaluation (Visual Analog Scale) | 1 year
  patient were asked to report the pain after the procedure in terms of visual analog scale (VAS) score in a rating between 1 to 10. There are 5-point verbal descriptive scale with an interval of 2("nil," "mild," "moderate," "severe," and "very severe") Patients were asked to rate their pain in a score between 1-10

CONTACTS AND LOCATIONS:
Overall Officials: PRIYANKA ACHARYA, mds, Principal Investigator — Rajiv Gandhi University of Health Sciences; prabhuji mlv, mds, Study Director — Rajiv Gandhi University of Health Sciences
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Trisi P, Berardini M, Falco A, Podaliri Vulpiani M. New Osseodensification Implant Site Preparation Method to Increase Bone Density in Low-Density Bone: In Vivo Evaluation in Sheep. Implant Dent. 2016 Feb;25(1):24-31. doi: 10.1097/ID.0000000000000358. PMID 26584202
- [Result] Lahens B, Neiva R, Tovar N, Alifarag AM, Jimbo R, Bonfante EA, Bowers MM, Cuppini M, Freitas H, Witek L, Coelho PG. Biomechanical and histologic basis of osseodensification drilling for endosteal implant placement in low density bone. An experimental study in sheep. J Mech Behav Biomed Mater. 2016 Oct;63:56-65. doi: 10.1016/j.jmbbm.2016.06.007. Epub 2016 Jun 10. PMID 27341291
- [Result] Lahens B, Lopez CD, Neiva RF, Bowers MM, Jimbo R, Bonfante EA, Morcos J, Witek L, Tovar N, Coelho PG. The effect of osseodensification drilling for endosteal implants with different surface treatments: A study in sheep. J Biomed Mater Res B Appl Biomater. 2019 Apr;107(3):615-623. doi: 10.1002/jbm.b.34154. Epub 2018 Aug 6. PMID 30080320
- [Result] Witek L, Neiva R, Alifarag A, Shahraki F, Sayah G, Tovar N, Lopez CD, Gil L, Coelho PG. Absence of Healing Impairment in Osteotomies Prepared via Osseodensification Drilling. Int J Periodontics Restorative Dent. 2019 Jan/Feb;39(1):65-71. doi: 10.11607/prd.3504. PMID 30543729
- [Result] Witek L, Alifarag AM, Tovar N, Lopez CD, Gil LF, Gorbonosov M, Hannan K, Neiva R, Coelho PG. Osteogenic parameters surrounding trabecular tantalum metal implants in osteotomies prepared via osseodensification drilling. Med Oral Patol Oral Cir Bucal. 2019 Nov 1;24(6):e764-e769. doi: 10.4317/medoral.23108. PMID 31655837
- [Result] Alifarag AM, Lopez CD, Neiva RF, Tovar N, Witek L, Coelho PG. Atemporal osseointegration: Early biomechanical stability through osseodensification. J Orthop Res. 2018 Sep;36(9):2516-2523. doi: 10.1002/jor.23893. Epub 2018 Mar 30. PMID 29537128
- [Result] Tian JH, Neiva R, Coelho PG, Witek L, Tovar NM, Lo IC, Gil LF, Torroni A. Alveolar Ridge Expansion: Comparison of Osseodensification and Conventional Osteotome Techniques. J Craniofac Surg. 2019 Mar/Apr;30(2):607-610. doi: 10.1097/SCS.0000000000004956. PMID 30507887
- [Result] Lopez CD, Alifarag AM, Torroni A, Tovar N, Diaz-Siso JR, Witek L, Rodriguez ED, Coelho PG. Osseodensification for enhancement of spinal surgical hardware fixation. J Mech Behav Biomed Mater. 2017 May;69:275-281. doi: 10.1016/j.jmbbm.2017.01.020. Epub 2017 Jan 13. PMID 28113132
- [Result] Huwais S, Meyer EG. A Novel Osseous Densification Approach in Implant Osteotomy Preparation to Increase Biomechanical Primary Stability, Bone Mineral Density, and Bone-to-Implant Contact. Int J Oral Maxillofac Implants. 2017 Jan/Feb;32(1):27-36. doi: 10.11607/jomi.4817. Epub 2016 Oct 14. PMID 27741329
- [Result] Stavropoulos A, Cochran D, Obrecht M, Pippenger BE, Dard M. Effect of Osteotomy Preparation on Osseointegration of Immediately Loaded, Tapered Dental Implants. Adv Dent Res. 2016 Mar;28(1):34-41. doi: 10.1177/0022034515624446. PMID 26927486
- [Result] Almutairi AS, Walid MA, Alkhodary MA. The effect of osseodensification and different thread designs on the dental implant primary stability. F1000Res. 2018 Dec 5;7:1898. doi: 10.12688/f1000research.17292.1. eCollection 2018. PMID 31131085
- [Result] Oliveira PGFP, Bergamo ETP, Neiva R, Bonfante EA, Witek L, Tovar N, Coelho PG. Osseodensification outperforms conventional implant subtractive instrumentation: A study in sheep. Mater Sci Eng C Mater Biol Appl. 2018 Sep 1;90:300-307. doi: 10.1016/j.msec.2018.04.051. Epub 2018 Apr 18. No abstract available. PMID 29853095
- [Result] Trisi P, Berardini M, Falco A, Podaliri Vulpiani M. Validation of value of actual micromotion as a direct measure of implant micromobility after healing (secondary implant stability). An in vivo histologic and biomechanical study. Clin Oral Implants Res. 2016 Nov;27(11):1423-1430. doi: 10.1111/clr.12756. Epub 2016 Jan 4. PMID 26727557
- [Result] Falco A, Berardini M, Trisi P. Correlation Between Implant Geometry, Implant Surface, Insertion Torque, and Primary Stability: In Vitro Biomechanical Analysis. Int J Oral Maxillofac Implants. 2018 Jul/Aug;33(4):824-830. doi: 10.11607/jomi.6285. PMID 30024998
- [Result] Slete FB, Olin P, Prasad H. Histomorphometric Comparison of 3 Osteotomy Techniques. Implant Dent. 2018 Aug;27(4):424-428. doi: 10.1097/ID.0000000000000767. PMID 29762184
- [Result] Cappare P, Vinci R, Di Stefano DA, Traini T, Pantaleo G, Gherlone EF, Gastaldi G. Correlation between Initial BIC and the Insertion Torque/Depth Integral Recorded with an Instantaneous Torque-Measuring Implant Motor: An in vivo Study. Clin Implant Dent Relat Res. 2015 Oct;17 Suppl 2:e613-20. doi: 10.1111/cid.12294. Epub 2015 Apr 15. PMID 25876078
- [Result] Alghamdi H, Anand PS, Anil S. Undersized implant site preparation to enhance primary implant stability in poor bone density: a prospective clinical study. J Oral Maxillofac Surg. 2011 Dec;69(12):e506-12. doi: 10.1016/j.joms.2011.08.007. PMID 22117707
- [Result] Markovic A, Calvo-Guirado JL, Lazic Z, Gomez-Moreno G, Calasan D, Guardia J, Colic S, Aguilar-Salvatierra A, Gacic B, Delgado-Ruiz R, Janjic B, Misic T. Evaluation of primary stability of self-tapping and non-self-tapping dental implants. A 12-week clinical study. Clin Implant Dent Relat Res. 2013 Jun;15(3):341-9. doi: 10.1111/j.1708-8208.2011.00415.x. Epub 2011 Dec 15. PMID 22171668